CLINICAL TRIAL: NCT04222101
Title: Association of Insulin Resistance and FGF21 on Cardiac Function in Pediatric Dilated Cardiomyopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Daniel Mak, MD, Principal Investigator, Le Bonheur Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19-06748-FB
Record Dates: First submitted 2019-12-19; First posted 2020-01-09 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Insulin Resistance
Keywords: pediatrics
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Insulin Resistance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cardiomyopathy (Other): only one arm, all participants undergo oral glucose tolerance testing and results are used to evaluate association with degree of cardiac dysfunction
  Interventions: Diagnostic Test: Oral glucose tolerance test

INTERVENTIONS:
Diagnostic Test: Oral glucose tolerance test — measure insulin, glucose and FGF21 levels in response to oral glucose challenge

SUMMARY:
This study will investigate whether there is an association between insulin resistance and cardiac function in children with dilated or hypertrophic cardiomyopathy. This study will also investigate whether there is an association between FGF21 and cardiac function in children with dilated or hypertrophic cardiomyopathy and whether this is mediated through greater insulin resistance and/or through independent effects.

DETAILED DESCRIPTION:
Although pediatric cardiomyopathy is rare, the condition is severe and life-threatening. The main focus of this proposed study will examine whether insulin resistance is correlated with decreased cardiac function which will hopefully pave the way for future clinical trials using medications that sensitize insulin such as metformin or glucagon-like peptide-1 (GLP-1 agonists) as possible therapeutic agents. The exploratory piece of this study will investigate a novel therapeutic target by determining whether FGF21 has any direct effects on cardiac function and whether it interacts with insulin resistance in altering cardiac function. Patients with cardiomyopathy normally undergo ECHO as part of routine evaluation and follow up and is standard of care. At this time, there are no official guidelines for pediatric patients with cardiomyopathy to undergo oral glucose tolerance testing (OGTT) and thus it is not part of the standard of care. Based on findings from this study, the investigators hope to justify performing an OGTT on pediatric patients with dilated or hypertrophic cardiomyopathy and incorporate the procedure in future practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dilated or hypertrophic cardiomyopathy
* Pubertal (Tanner 2 breast in females or testicular volume ≥ 4mL in males)
* Permission by the primary cardiologist of the patient for enrollment in the study

Exclusion Criteria:

* Prior diagnosis of diabetes and treatment with anti-diabetes medication
* Neuromuscular disorder
* Inborn error of metabolism
* Malformation syndrome
* Clinically unstable based on the assessment of the primary cardiologist caring for the patient
* inability of parent/legal guardian to provide informed consent
* non-English speaking

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Whole body insulin sensitivity index | baseline
  correlate whole body insulin sensitivity index with left ventricular ejection fraction

SECONDARY OUTCOMES:
FGF21 level | baseline
  correlate FGF21 levels with whole body sensitivity index and left ventricular ejection fraction

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Mak, MD, Principal Investigator — Le Bonheur/UTHSC Pediatric Endocrine fellowship
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a single center, pilot study; data will not be made available but findings from the study will be published

REFERENCES:
- [Background] Towbin JA, Lowe AM, Colan SD, Sleeper LA, Orav EJ, Clunie S, Messere J, Cox GF, Lurie PR, Hsu D, Canter C, Wilkinson JD, Lipshultz SE. Incidence, causes, and outcomes of dilated cardiomyopathy in children. JAMA. 2006 Oct 18;296(15):1867-76. doi: 10.1001/jama.296.15.1867. PMID 17047217
- [Background] Neglia D, De Caterina A, Marraccini P, Natali A, Ciardetti M, Vecoli C, Gastaldelli A, Ciociaro D, Pellegrini P, Testa R, Menichetti L, L'Abbate A, Stanley WC, Recchia FA. Impaired myocardial metabolic reserve and substrate selection flexibility during stress in patients with idiopathic dilated cardiomyopathy. Am J Physiol Heart Circ Physiol. 2007 Dec;293(6):H3270-8. doi: 10.1152/ajpheart.00887.2007. Epub 2007 Oct 5. PMID 17921325
- [Background] Riehle C, Abel ED. Insulin Signaling and Heart Failure. Circ Res. 2016 Apr 1;118(7):1151-69. doi: 10.1161/CIRCRESAHA.116.306206. PMID 27034277
- [Background] Fisher FM, Maratos-Flier E. Understanding the Physiology of FGF21. Annu Rev Physiol. 2016;78:223-41. doi: 10.1146/annurev-physiol-021115-105339. Epub 2015 Nov 19. PMID 26654352
- [Background] Camporez JP, Jornayvaz FR, Petersen MC, Pesta D, Guigni BA, Serr J, Zhang D, Kahn M, Samuel VT, Jurczak MJ, Shulman GI. Cellular mechanisms by which FGF21 improves insulin sensitivity in male mice. Endocrinology. 2013 Sep;154(9):3099-109. doi: 10.1210/en.2013-1191. Epub 2013 Jun 13. PMID 23766126
- [Result] Shah A, Shannon RP. Insulin resistance in dilated cardiomyopathy. Rev Cardiovasc Med. 2003;4 Suppl 6:S50-7. PMID 14668703
- [Result] Davila-Roman VG, Vedala G, Herrero P, de las Fuentes L, Rogers JG, Kelly DP, Gropler RJ. Altered myocardial fatty acid and glucose metabolism in idiopathic dilated cardiomyopathy. J Am Coll Cardiol. 2002 Jul 17;40(2):271-7. doi: 10.1016/s0735-1097(02)01967-8. PMID 12106931
- [Result] Nikolaidis LA, Sturzu A, Stolarski C, Elahi D, Shen YT, Shannon RP. The development of myocardial insulin resistance in conscious dogs with advanced dilated cardiomyopathy. Cardiovasc Res. 2004 Feb 1;61(2):297-306. doi: 10.1016/j.cardiores.2003.11.027. PMID 14736546
- [Result] Swan JW, Anker SD, Walton C, Godsland IF, Clark AL, Leyva F, Stevenson JC, Coats AJ. Insulin resistance in chronic heart failure: relation to severity and etiology of heart failure. J Am Coll Cardiol. 1997 Aug;30(2):527-32. doi: 10.1016/s0735-1097(97)00185-x. PMID 9247528
- [Result] Witteles RM, Tang WH, Jamali AH, Chu JW, Reaven GM, Fowler MB. Insulin resistance in idiopathic dilated cardiomyopathy: a possible etiologic link. J Am Coll Cardiol. 2004 Jul 7;44(1):78-81. doi: 10.1016/j.jacc.2004.03.037. PMID 15234411
- [Result] Sakai Y, Maruyama T, Katsuta H, Kogawa K, Akashi T, Izumi K, Tominaga H, Kono S, Nagafuchi S, Harada M. Patients with dilated cardiomyopathy possess insulin resistance independently of cardiac dysfunction or serum tumor necrosis factor-alpha. Int Heart J. 2006 Nov;47(6):877-87. doi: 10.1536/ihj.47.877. PMID 17268122